CLINICAL TRIAL: NCT00777699
Title: A Phase 1 Dose-Escalation Study of XL765 in Combination With Erlotinib in Subjects With Solid Tumors
Brief Title: Safety Study of XL765 (SAR245409) in Combination With Erlotinib in Adults With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED11442; 2008-003219-11 (EudraCT Number); XL765-003 (Other: (other study code))
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Cancer; Non-Small Cell Lung Cancer
Keywords: Cancer; Solid Tumors; NSCLC
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — XL765; Erlotinib Hydrochloride

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: XL765 (SAR245409); Drug: erlotinib

INTERVENTIONS:
Drug: XL765 (SAR245409) — Gelatin capsules supplied in 5-mg, 10-mg, and 50-mg strengths; daily dosing
Drug: erlotinib — Tablets supplied in 25-mg, 100-mg, and 150-mg strengths; daily dosing
  Other Names: Tarceva®

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of XL765 in combination with erlotinib (Tarceva®) in subjects with solid tumors. XL765 is a new chemical entity that inhibits the kinases PI3K and mTOR. In preclinical studies, inactivation of PI3K has been shown to inhibit growth and induce apoptosis (programmed cell death) in tumor cells, whereas inactivation of mTOR has been shown to inhibit the growth of tumor cells. Erlotinib is an orally administered inhibitor of EGFR (also known as HER1) tyrosine kinase. It was approved by the FDA as a single agent for the treatment of patients with locally advanced or metastatic non-small-cell lung cancer (NSCLC) after failure of at least one prior chemotherapy regimen and in combination with gemcitabine for first line treatment of patients with locally advanced, unresectable or metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of:

  * Advanced solid tumor that is no longer responding to therapies OR
  * Advanced or metastatic NSCLC that has previously been treated with erlotinib or gefitinib
* ECOG Performance Status 0-1
* Adequate organ and bone arrow function as defined by hematological and serum chemistry limits
* At least 18 years old
* Both men and women must practice adequate contraception
* Informed consent

Exclusion Criteria:

* Restriction of some therapies/medications within specific timeframes prior to enrollment and during the study including prior therapy with PI3K, cytotoxic chemotherapy, biologic agents, nitrosoureas or mitomycin C, small-molecule kinase inhibitors, non-cytotoxic hormonal agents
* Erlotinib intolerant
* Taking oral corticosteroids chronically or > 1 mg/day warfarin
* Not recovered from the toxic effects of prior therapy
* History of diabetes mellitus and an HgbA1c > 7%
* Uncontrolled intercurrent illness
* Pregnant or breastfeeding
* Congestive heart failure, unstable angina, or a myocardial infarction within 3 months of entering the study.
* HIV positive
* Diagnosis of another malignancy may exclude subject from study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability, and maximum tolerated dose of XL765 administered in combination with erlotinib | Assessed during periodic visits

SECONDARY OUTCOMES:
To evaluate plasma pharmacokinetics of XL765 and erlotinib when administered in combination | Assessed during periodic visits
To evaluate preliminary efficacy of XL765 in combination with erlotinib in subjects with non-small-cell lung cancer (NSCLC) and other solid tumors | Assessed during periodic visits

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 168983, Philadelphia, Pennsylvania, United States